CLINICAL TRIAL: NCT02166762
Title: Mapping of the Coronary Venous System in Patients With Heart Failure Presenting for CRT-D (Cardiac Resynchronization Therapy) Implantation. Correlating QLV Interval to Fluoroscopic LV (Left Ventricular) Lead Position.
Brief Title: Correlating QLV Interval to Left Ventricular (LV) Lead Position in Patients Receiving Cardiac Resynchronization Therapy.
Acronym: QLV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Ulrika Birgersdotter-Green, Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121099
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure; Cardiomyopathy; Cardiac Arrhythmia
Keywords: Cardiac Resynchronization Therapy; Biventricular implantable cardioverter defibrillators; Heart failure; Cardiomyopathy; QLV; LV lead placement; Arrhythmia
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QLV interval measurement (Experimental): QLV measurements collected during implantation of CRT-D device
  Interventions: Procedure: QLV interval measurement

INTERVENTIONS:
Procedure: QLV interval measurement — Measurements of the QLV interval is defined from the onset of the QRS width of the surface ECG to the first large positive or negative peak of the LV EGM during a cardiac cycle. Recorded EGM's will be measured at three distinct points (basal, mid, and distal) within each target vessel.

SUMMARY:
This is a prospective clinical trial to determine the optimal QLV interval during implantation to achieve the best possible response from cardiac resynchronization therapy for heart failure patients.

DETAILED DESCRIPTION:
Heart failure is a growing epidemic in the United States. Heart failure is associated with shortness of breath, reduced exercise tolerance, and manifestations of peripheral fluid retention. As the disease progresses, there is development of cardiac dyssynchrony (failure of the heart to act as one unit) in the electrical and mechanical functions of the myocardium.

During implantation of a cardiac resynchronization therapy defibrillator (CRT-D) device, three electrical wires are placed in the right atrium (RA), right ventricle (RV) and coronary venous system that drains blood from the left ventricle (LV). The LV lead is placed in the posterolateral tributaries of the coronary venous system using special delivery tools. Pacing therapies to resynchronize the heart have been shown to improve functional class and mortality in patients with severe heart failure i.e. New York Heart Association (NYHA) class III and IV functional status. Current indications for cardiac resynchronization therapy (CRT-D) include severe cardiomyopathy (Ejection Fraction < 35%), with shortness of breath at rest or minimal exertion (NYHA class II, IV), prolonged QRS > 130ms on surface echocardiogram (ECG) and life expectancy more than one year. CRT-D therapy results in decrease of heart failure admissions and improvements in quality of life.

Response to CRT is associated with improvement in functional status by one NYHA functional class schema or by evidence of reverse remodeling (decrease in end systolic LV dimension by 15%). However across clinical trials, a third of the patients are non-responders to CRT therapy. Non-ischemic etiology of heart failure and presence of electrical dyssynchrony on surface ECG suggested by QRS >150ms are associated with better response with CRT. Non response to CRT can be due to inappropriate patient selection, inappropriate device programming, and inappropriate lead placement. However, inappropriate lead placement is the factor that can be changed during device implantation. Adverse changes in morality and heart failure can occur with sub-optimal position of the LV lead. Most echocardiographic parameters to predict responders were not clinically useful. Appropriate positioning near the area of the heart with latest activation (usually posterolateral segment of the left ventricle) is associated with better response. Inter-ventricular delay as measured by the time delay between the two leads in the left and right ventricles (RV-LV delay) was shown to be a better predictor of response. Interval from the first deflection of the surface ECG to the bipolar electrogram (QLV interval) can be used as a surrogate to identify the delayed segments of the left ventricle. Preliminary studies have shown better response using this approach of lead placement in the regions of latest activation. SMART AV study which used a similar algorithm in assessing delay also showed a trend for better response using QLV interval. However, the fluoroscopic lead position was not correlated with QLV interval for that study. We plan to measure this area of delayed activation to target effective lead placement and map the coronary veins to target the longest QLV interval in each patient.

For this study, medical history and demographic information will be collected from patients as well as clinical information from the procedure. The QLV measurements will be collected prior to implant of LV lead. The QLV interval is defined as the measurement from the onset of the QRS width of the surface ECG to the first large positive or negative peak of the LV electrogram (EGM) during a cardiac cycle. QLV EGM will be taken from either the LV pacing lead and/or .014 wire. QLV EGM's will be measured at three distinct points (basal, mid, and distal) within each target vessel. Each data point will be the average of four to six beats to allow for respiratory variance, and recorded using the Bard mapping system. The final lead position will be the area of vein that has the longest QLV interval with appropriate sensing and pacing thresholds. The QLV measurements will be conducted, in addition to all standard of care procedures for CRT-D implantation for patients enrolled in the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are indicated for CRT-D devices according to the current guidelines for implantation of cardiac pacemakers and antiarrhythmia devices

Exclusion Criteria:

* Patients who are under the age of 18
* Patients who are pregnant
* Patients who cannot have intravenous contrast due to allergic reactions or chronic renal insufficiency
* Patients who are unable or unwilling for any reason to consent for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
QLV measurement | 15 minutes
  Measurements of the QLV interval is defined from the onset of the QRS width of the surface ECG to the first large positive or negative peak of the LV electrogram (EGM) during a cardiac cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Birgersdotter-Green, MD, Principal Investigator — UCSD Electrophysiology
Locations (1):
- UCSD Sulpizio Cardiovascular Center, La Jolla, California, United States

REFERENCES:
- [Background] McAlister FA, Ezekowitz J, Hooton N, Vandermeer B, Spooner C, Dryden DM, Page RL, Hlatky MA, Rowe BH. Cardiac resynchronization therapy for patients with left ventricular systolic dysfunction: a systematic review. JAMA. 2007 Jun 13;297(22):2502-14. doi: 10.1001/jama.297.22.2502. PMID 17565085
- [Background] Epstein AE, Dimarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO; American College of Cardiology/American Heart Association Task Force on Practice; American Association for Thoracic Surgery; Society of Thoracic Surgeons. ACC/AHA/HRS 2008 guidelines for Device-Based Therapy of Cardiac Rhythm Abnormalities: executive summary. Heart Rhythm. 2008 Jun;5(6):934-55. doi: 10.1016/j.hrthm.2008.04.015. Epub 2008 May 19. No abstract available. PMID 18534377
- [Background] Feldman AM, de Lissovoy G, Bristow MR, Saxon LA, De Marco T, Kass DA, Boehmer J, Singh S, Whellan DJ, Carson P, Boscoe A, Baker TM, Gunderman MR. Cost effectiveness of cardiac resynchronization therapy in the Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) trial. J Am Coll Cardiol. 2005 Dec 20;46(12):2311-21. doi: 10.1016/j.jacc.2005.08.033. PMID 16360064
- [Background] Singh JP, Klein HU, Huang DT, Reek S, Kuniss M, Quesada A, Barsheshet A, Cannom D, Goldenberg I, McNitt S, Daubert JP, Zareba W, Moss AJ. Left ventricular lead position and clinical outcome in the multicenter automatic defibrillator implantation trial-cardiac resynchronization therapy (MADIT-CRT) trial. Circulation. 2011 Mar 22;123(11):1159-66. doi: 10.1161/CIRCULATIONAHA.110.000646. Epub 2011 Mar 7. PMID 21382893
- [Background] Chung ES, Leon AR, Tavazzi L, Sun JP, Nihoyannopoulos P, Merlino J, Abraham WT, Ghio S, Leclercq C, Bax JJ, Yu CM, Gorcsan J 3rd, St John Sutton M, De Sutter J, Murillo J. Results of the Predictors of Response to CRT (PROSPECT) trial. Circulation. 2008 May 20;117(20):2608-16. doi: 10.1161/CIRCULATIONAHA.107.743120. Epub 2008 May 5. PMID 18458170
- [Background] Butter C, Auricchio A, Stellbrink C, Fleck E, Ding J, Yu Y, Huvelle E, Spinelli J; Pacing Therapy for Chronic Heart Failure II Study Group. Effect of resynchronization therapy stimulation site on the systolic function of heart failure patients. Circulation. 2001 Dec 18;104(25):3026-9. doi: 10.1161/hc5001.102229. PMID 11748094
- [Background] Singh JP, Fan D, Heist EK, Alabiad CR, Taub C, Reddy V, Mansour M, Picard MH, Ruskin JN, Mela T. Left ventricular lead electrical delay predicts response to cardiac resynchronization therapy. Heart Rhythm. 2006 Nov;3(11):1285-92. doi: 10.1016/j.hrthm.2006.07.034. Epub 2006 Aug 10. PMID 17074633
- [Background] Gold MR, Niazi I, Giudici M, Leman RB, Sturdivant JL, Kim MH, Yu Y, Ding J, Waggoner AD. A prospective comparison of AV delay programming methods for hemodynamic optimization during cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2007 May;18(5):490-6. doi: 10.1111/j.1540-8167.2007.00770.x. Epub 2007 Feb 21. PMID 17313533
- [Background] Khan FZ, Virdee MS, Palmer CR, Pugh PJ, O'Halloran D, Elsik M, Read PA, Begley D, Fynn SP, Dutka DP. Targeted left ventricular lead placement to guide cardiac resynchronization therapy: the TARGET study: a randomized, controlled trial. J Am Coll Cardiol. 2012 Apr 24;59(17):1509-18. doi: 10.1016/j.jacc.2011.12.030. Epub 2012 Mar 7. PMID 22405632
- [Background] Ellenbogen KA, Gold MR, Meyer TE, Fernndez Lozano I, Mittal S, Waggoner AD, Lemke B, Singh JP, Spinale FG, Van Eyk JE, Whitehill J, Weiner S, Bedi M, Rapkin J, Stein KM. Primary results from the SmartDelay determined AV optimization: a comparison to other AV delay methods used in cardiac resynchronization therapy (SMART-AV) trial: a randomized trial comparing empirical, echocardiography-guided, and algorithmic atrioventricular delay programming in cardiac resynchronization therapy. Circulation. 2010 Dec 21;122(25):2660-8. doi: 10.1161/CIRCULATIONAHA.110.992552. Epub 2010 Nov 15. PMID 21098426